CLINICAL TRIAL: NCT02450773
Title: Furosemide for Prevention of Severe Postpartum Hypertension: a Randomized Controlled Trial
Brief Title: Prevention of Severe Postpartum Hypertension
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, Professor of Obstetrics and Gynecology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201501157
Record Dates: First submitted 2015-05-11; First posted 2015-05-21 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: postpartum; preeclampsia; gestational hypertension
MeSH Terms: conditions — Hypertension; Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Furosemide; Potassium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide/Potassium chloride (Experimental): 40 mg furosemide; 20 meq potassium chloride
  Interventions: Drug: Furosemide; Drug: Potassium chloride
- Placebo (Placebo Comparator): Placebo #1, Placebo #2
  Interventions: Drug: Placebo #1; Drug: Placebo #2

INTERVENTIONS:
Drug: Furosemide — 40 mg furosemide on postpartum day 1-6
  Other Names: Lasix
  Arms: Furosemide/Potassium chloride
Drug: Potassium chloride — 20 meq potassium chloride on postpartum day 1-6
  Other Names: KCl
  Arms: Furosemide/Potassium chloride
Drug: Placebo #1 — Placebo (for furosemide)
  Arms: Placebo
Drug: Placebo #2 — Placebo (for KCl)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether postpartum administration of furosemide to women with antepartum hypertensive disorders (gestational hypertension, preeclampsia) or elevated blood pressure in the first 24 hours following delivery reduces severe postpartum hypertension.

ELIGIBILITY:
Inclusion Criteria:

Women > 18 years of age or emancipated minors

Women undergoing vaginal or cesarean delivery at > 23 weeks gestation with:

* Antepartum diagnosis of gestational hypertension
* Antepartum diagnosis of preeclampsia
* Antepartum diagnosis of preeclampsia with severe features
* Mild hypertension (<150/100) in first 24 hours following delivery

Exclusion Criteria:

* Chronic hypertension
* Allergy to furosemide
* Pre-existing hypokalemia (serum K < 3.0 meq/L)
* Chronic kidney disease
* Serum Cr > 1.1
* Inability to obtain informed consent
* Pre-existing diuretic use
* Oliguria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Composite maternal morbidity | 0-6 weeks following delivery
  Requiring antihypertensive medication at discharge, readmission for blood pressure, end-organ damage from hypertension

SECONDARY OUTCOMES:
Adverse events associated with furosemide | 0-6 weeks following delivery
  Hypokalemia
Adverse events associated with furosemide | 0-6 weeks following delivery
  hyperglycemia
Adverse events associated with furosemide | 0-6 weeks following delivery
  oliguria
Adverse events associated with furosemide | 0-6 weeks following delivery
  hypotension
Adverse events associated with furosemide | 0-6 weeks following delivery
  elevated serum creatinine

OTHER OUTCOMES:
Cardiovascular changes following delivery | 0-1 week following delivery
  Maternal echocardiogram, renin, aldosterone, B-natriuretic peptide levels

CONTACTS AND LOCATIONS:
Overall Officials: Methodius G Tuuli, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri